CLINICAL TRIAL: NCT03358368
Title: A Prospective Single-centre Pilot Study to Assess a Magnetocardiograph Device in Patients Following Myocardial Infarction.
Brief Title: MCG Post Myocardial Infarction Study
Status: Completed | Type: Observational
Sponsor: Creavo Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP 004
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vitalscan — Vitalscan is a magnetocardiograph device

SUMMARY:
The study is being performed to evaluate a new portable medical device, the Creavo Vitalscan Magnetocardiograph (Vitalscan) on patients who have had a confirmed myocardial infarction (heart attack) within the previous 12 weeks.

DETAILED DESCRIPTION:
Magnetocardiography (MCG) is a non-contact, passive, imaging technique that detects the magnetic fields generated by the electrical activity of the heart. The MCG technology has been evaluated in several clinical studies, demonstrating its potential usefulness in the detection of patients with stable angina and acute coronary syndrome (ACS), including non-ST segment elevation myocardial infarction (NSTEMI).

Previous studies have been completed using earlier versions of the Vitalscan device. Results showed that the device could differentiate between patients with confirmed ischaemic heart disease (IHD) and NSTEMI, those with non-IHD experiencing chest pain and healthy (non-ischaemic) control subjects.

The aim of this pilot study is to assess the difference between abnormal MCG images from patients with a confirmed and recent myocardial infarction (MI)and normal images from previously obtained healthy volunteer controls scanned with the current device, so that comparisons can be made to the data acquired from the previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed myocardial infarction within 12 weeks of the initial event
* Patients admitted to the Coronary Care Unit (CCU) at Warwick Hospital on the point of discharge or patients already discharged from the CCU attending the cardiac rehabilitation classes
* 18+ year old male or female
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* Atrial fibrillation
* Thoracic metal implants (cardiac stents allowed)
* Pacemaker or internal defibrillator
* Pregnancy (if after 20-week period)* or lactation
* Patient unable to lie down (i.e. supine position up to a maximum 25 degree tilt) or stay still on the examination bed
* Patient unable to understand the informed consent process and/or has a poor understanding of English (e.g. English-speaking relative/translator not available)

  * There should not be any effect on pregnancy due to the non-invasive nature of the device. Pregnancy after the 20-week period excluded from the study due to the size and position of the foetus and unknown possibility of picking up the foetal heartbeat, rendering the scan non-usable for study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a confirmed myocardial infarction within 12 weeks of the initial event under the care of South Warwickshire NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
MCG parameter extraction | From baseline scan
  To extract parameters from MCG scans to identify key characteristics (markers) for myocardial infarction

SECONDARY OUTCOMES:
MCG parameter analysis | From baseline scan
  To use the markers identified to differentiate between abnormal (post MI) images and normal (healthy volunteer) images using evaluation performance measures

CONTACTS AND LOCATIONS:
Overall Officials: Roger Beadle, MBBS, Principal Investigator — South Warwickshire NHS Foundation Trust, UK
Locations (1):
- South Warwickshire NHS Trust, Warwick, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No